CLINICAL TRIAL: NCT07214337
Title: Feasibility, Adoption and Efficacy of Digital Inhaler in the Management of Obstructive Lung Disease
Brief Title: Digital Inhaler Use in Obstructive Lung Disease Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Breathe California, Los Angeles County (Other)
Responsible Party: Principal Investigator, Sara Ghandehari, Professor of Medicine, Division of Pulmonary and Critical Care Medicine, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00004080
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Obstructive Airways Disease Exacerbated; Chronic Obstructive Airway Disease
Keywords: Chronic Obstructive Airways Disease; COPD; COPD Exacerbation; Severe COPD; Moderate COPD; Severe Chronic Obstructive Airways Disease; Moderate Chronic Obstructive Airways Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Digital Inhaler Attachment for Regular Care (Other): This group of patients will be provided interactive device that provides inhaler coaching for to use for 6 month duration.
  Interventions: Device: Digital Inhaler Attachment

INTERVENTIONS:
Device: Digital Inhaler Attachment — This intervention is the attachment of a digital device to provide patient with coaching for optimal inhaler use and technique, as well as monitoring of patient use of inhaler to patient and health care team. Patient will continue to use inhalers prescribed as per usual care for management of COPD.

SUMMARY:
This is a pilot study to evaluate the role digital inhaler technology on patients with obstructive lung disease in preventing admissions and exacerbation, as well as improving symptom control. The primary objective is to evaluate feasibility of study protocol, patient recruitment, and patient retention with goal recruitment of 20 participants, 60% recruitment success, and 60% retention rate for 6 months duration. The secondary objectives are the evaluation of patient admission rate, exacerbation rates, and symptoms control with use of digital inhaler technology The subject population will be patients with physician diagnosed obstructive lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Any sex
* Over the age of 18 years.
* Physician-diagnosed obstructive lung disease
* Speak, read, and understand English.
* The current study is a feasibility pilot. Based on the results of the study, future studies will include non-English speakers as well.
* Able to understand study requirements and comply with study procedures.
* Ability to operate a smartphone or tablet (for questionnaire and symptoms input).
* Patients who use either a DPI or an MDI device as controller medications. Medications will not be changed by the study team.

Exclusion Criteria:

* Physically disabled such that they are incapable of using digital devices or metered dose inhalers.
* Suffer from any visual, hearing or cognitive impairment that cannot be corrected enough to operate the devices properly. Mild/moderate vision loss and mild hearing loss may be included with appropriate corrective measures that do not affect the device usage.
* Suffering from serious uncontrolled medical conditions that may interfere with study conduct.
* Inability or unwillingness of the participant to give written informed consent.
* Pregnant women (due to complicated physiology)
* The current study is a feasibility pilot. Based on the results of the study, future studies will likely include pregnant patients as well.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment Percentage | 6 months
  The investigators will be looking at what percentage of patients approached for recruitment choose to participate in the study. Accrual rate will be computed as the proportion of subjects enrolled as a function of the number of subjects screened.
Participant Retention Percentage | 6 months
  The investigators will also be looking at what percentage patient who choose to participate remain participating for the full 6-month duration of the study period. The retention rate over the full 6-month period of follow-up will be computed among enrolled subjects.

SECONDARY OUTCOMES:
Re-admission Rate | 6 months
  Hospital re-admission rate for COPD exacerbation during study period
COPD Exacerbation Rates | 6 months
  Rates of COPD exacerbation after intervention during study period
Symptom Control | 6 months
  Overall symptoms control of COPD after intervention during study period. This will utilize the COPD Assessment Test. Scores with this test can range from 0 to 40, with higher score representing worse severity of disease and worse symptom control.
Satisfaction with Device Assessed with Questionnaire | 6 months
  Assessment of patient satisfaction with use of device utilizing questionnaire to be administered at the conclusion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ghandehari, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.lung.org/research/trends-in-lung-disease/copd-trends-brief/copd-mortality
- See also: Related Info — https://www.lung.org/research/trends-in-lung-disease/copd-trends-brief/copd-prevalence
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/chronic-obstructive-pulmonary-disease-(copd)
- See also: Related Info — https://www.nature.com/articles/pcrj201375